CLINICAL TRIAL: NCT03049969
Title: Cognitive Remediation Augmented With Transcranial Direct Current Stimulation (tDCS)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: New controlled trial was funded, this study was no longer needed.
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-01810
Record Dates: First submitted 2017-02-08; First posted 2017-02-10 (Actual); Results first posted 2024-06-18 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-06

CONDITIONS: Multiple Sclerosis; Neurological Disorder
Keywords: Working Memory; Cognitive Training; Transcranial Magnetic Stimulation
MeSH Terms: conditions — Multiple Sclerosis; Nervous System Diseases | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: 20 sessions of cognitive remediation while receiving 20 minutes of up to 2.0 mA tDCS using a DLPFC montage
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Cognitive Remediation (Experimental): For the 20 cognitive remediation sessions, eligible participants will receive 20 minutes of active tDCS stimulation (up to 2.0 mA, dorsolateral prefrontal cortex (dlPFC) motage) while they complete the cognitive training tasks. Once the participant has completed his/her 20 sessions a pre/post treatment assessment measures will be completed.
  Interventions: Device: tDCS stimulation

INTERVENTIONS:
Device: tDCS stimulation — up to 4.0 mA, dorsolateral prefrontal cortex (montage dependent on specific area of deficit) while completing cognitive training tasks
  Other Names: Soterix Mini-CT

SUMMARY:
The proposed study will test the feasibility and tolerability of transcranial direct current stimulation (tDCS) added to a cognitive remediation program in n=100 adults. For 60 cognitive remediation sessions, participants will receive 20 minutes of active tDCS stimulation (up to 4.0 mA, dorsolateral prefrontal cortex or montage dependent on specific area of deficit) while they complete the cognitive training tasks.

DETAILED DESCRIPTION:
Transcranial Direct Current Stimulation (tDCS) is a novel, safe, well-tolerated, and low-cost treatment approach that may enhance the benefits of cognitive remediation. The application of tDCS is a relatively recent therapeutic development that utilizes low amplitude direct currents to induce changes in cortical excitability. To meet this study's objectives, investigators will focus specifically on working memory (WM) in both training and outcome. Limiting training to WM exercises will provide the opportunity to test proof of concept for the combined therapies within this shorter two-week time frame, and maximize the synergistic effect by engaging the same regions as targeted by the tDCS.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Clinician Referral for cognitive remediation.
* Have undergone a neurological examination and neuropsychological examination as part of standard of care.
* Has access to internet service at home compatible with the study laptop (Wi-Fi or ethernet cable)
* Able to commit to the designated period of study training sessions with baseline and follow-up visits.
* Able to understand the informed consent process and provide consent to participate in the study

Exclusion Criteria:

* Visual, auditory and motor deficits that would prevent full ability to understand study instructions or operate the tDCS device or study laptop, as judged by treating clinician or study staff
* Primary, uncontrolled psychiatric disorder that would influence ability to participate
* Poorly controlled epilepsy
* Medical device implanted in the head (such as Deep Brain Stimulator) or in the neck (such as a Vagus Nerve Stimulator)
* Any skin disorder/sensitive skin (e.g., eczema, severe rashes), blisters, open wounds, burn including sunburns, cuts or irritation, or other skin defects which compromise the integrity of the skin at or near stimulation locations (where electrodes are placed)
* Treatment for a communicable skin disorder currently or over the past 12 months
* Other serious uncontrolled medical condition (e.g., cancer or acute myocardial infarction)
* Wide Range Achievement Test-4th Edition (WRAT-4) Reading Recognition score <85*
* Symbol Digit Modalities Test (SDMT) ≥3.0 SD below published norms*
* Learned English language after 12 years of age
* Pregnant or breastfeeding

  * In the case of the potential participant having either speech, motor or vision impairment secondary to their condition that will limit the completion of the SDMT and WRAT-4 screening measures the substitutions as mentioned above will be used.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-02-07 (Actual); Primary Completion 2023-03-26 (Actual); Study Completion 2023-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leigh Charvet, MD, Principal Investigator — New York University Medical Center Institutional Review Boards
Locations (1):
- New York University Medical Center, New York, New York, United States

REFERENCES:
- [Derived] Pilloni G, Shaw M, Feinberg C, Clayton A, Palmeri M, Datta A, Charvet LE. Long term at-home treatment with transcranial direct current stimulation (tDCS) improves symptoms of cerebellar ataxia: a case report. J Neuroeng Rehabil. 2019 Mar 19;16(1):41. doi: 10.1186/s12984-019-0514-z. PMID 30890162

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cognitive Remediation
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cognitive Remediation
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.33 (17.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 5
  More than one race | 0
  Unknown or Not Reported | 8
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Completing at Least 80% of the Targeted Number of Sessions.
Description: The protocol is designed to have a decision-tree series of checkpoints that must be met in order to proceed at each step
Time Frame: End of treatment (up to 12 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Cognitive Remediation
Number analyzed (Participants) | 15
Participants | 10

2. Primary Outcome: Number of Participants With Treatment Related Adverse Events
Time Frame: End of treatment (up to 12 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Cognitive Remediation
Number analyzed (Participants) | 15
Participants | 14

3. Secondary Outcome: Change in Visual Analogue Scale (VAS) for Pain Score
Description: VAS is a tool widely used to measure pain. A patient is asked to indicate his/her perceived pain intensity (most commonly) along a 10 mm horizontal line, and this rating is then measured from the left edge (=VAS score). The total score range is 0 (no pain) to 10 (worst pain imaginable); the higher the score, the worse the pain.
Time Frame: Baseline, end of treatment (up to 12 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Remediation
Number analyzed (Participants) | 12
score on a scale | -1.17 (5.37)

4. Secondary Outcome: Change in Negative Affect Score From the Positive and Negative Affect Scale (PANAS)
Description: This brief scale is comprised of 10 items measuring negative affect (e.g., upset, afraid). Individual items are scored 1-5, 1 being "very slightly or not at all" and 5 being "Extremely". The negative affect score is calculated by finding the sum of the 10 negative items. Scores range from 10 - 50. For the total negative score, a lower score indicates less of a negative affect.
Time Frame: Baseline, end of treatment (up to 12 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Remediation
Number analyzed (Participants) | 11
score on a scale | -3 (5.74)

5. Secondary Outcome: Change in Positive Affect Score From the Positive and Negative Affect Scale (PANAS)
Description: This brief scale is comprised of 10 items measuring positive affect (e.g., excited, inspired). Individual items are scored 1-5, 1 being "very slightly or not at all" and 5 being "Extremely". The positive affect score is calculated by finding the sum of the 10 positive items. Scores range from 10 - 50. For the total positive score, a higher score indicates more of a positive affect.
Time Frame: Baseline, end of treatment (up to 12 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Remediation
Number analyzed (Participants) | 12
score on a scale | -1.17 (5.37)

6. Secondary Outcome: Change in Symbol Digit Modalities Test (SDMT) Score
Description: The SDMT is a cognitive processing speed test. Participants are given a key of nine symbol-digit pairs along with a sequence of symbols. They are then asked to use the key to match as many symbols in the sequence to their corresponding numbers as possible within 90 seconds. The score is the number of correctly coded items from 0-110 in 90 seconds. Lower scores indicate cognitive decline.
Time Frame: Baseline, end of treatment (up to 12 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Remediation
Number analyzed (Participants) | 8
score on a scale | 0.75 (4.56)

ADVERSE EVENTS:
Time Frame: 12 Weeks
Arm/Group | Cognitive Remediation
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 14/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cognitive Remediation (N=15)
Tingling Sensation (Skin and subcutaneous tissue disorders) | 14
Itching Sensation (Skin and subcutaneous tissue disorders) | 14
Warmth Sensation (Skin and subcutaneous tissue disorders) | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-30): https://cdn.clinicaltrials.gov/large-docs/69/NCT03049969/Prot_SAP_000.pdf